CLINICAL TRIAL: NCT07274865
Title: Prevalence of Psychiatric Problems Among Patients and Healthcare Providers in the Department of Cardiovascular Medicine
Brief Title: Prevalence of Psychiatric Problems Among Patients and Healthcare Providers in a Cardiology Department: A Cross-Sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Loly Abdulhameed Abdullah, dr, Assiut University
Other Study IDs: psychiatry in cardiology
Record Dates: First submitted 2025-09-25; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Anxiety Depression; Burnout; Sleep
Keywords: psychiatric probldems in cardiologists; psychiatric problems in cardiovascular patients
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psychological Assessment using Validated Questionnaires — Participants will complete validated mental health questionnaires, including SCL-90R, COPE Inventory, Eysenck Personality Questionnaire, Perceived Stress Scale (PSS), Pittsburgh Sleep Quality Index (PSQI). Healthcare providers will additionally complete the Maslach Burnout Inventory (MBI). No experimental treatment or behavioral intervention will be applied.

SUMMARY:
The goal of this observational cross-sectional study is to determine the prevalence of psychiatric problems (depression, anxiety, stress, and burnout) among patients with cardiovascular diseases and healthcare providers working in the Department of Cardiovascular Medicine at Assiut University Heart Hospital.

The main questions it aims to answer are:

* What is the prevalence of depression, anxiety, and stress among cardiovascular patients?
* What is the prevalence of burnout, depression, and anxiety among healthcare providers in the same department?

The study will also explore potential sociodemographic, occupational, and clinical factors associated with these psychological outcomes.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVDs) remain the leading cause of morbidity and mortality worldwide. Psychological comorbidities-such as depression, anxiety, post-traumatic stress disorder, and cognitive impairment-are highly prevalent among patients with CVD and are known to adversely affect treatment adherence, quality of life, and overall outcomes.

Similarly, healthcare professionals working in cardiovascular medicine are exposed to continuous psychological stress due to long working hours, critical decision-making, and frequent exposure to life-threatening situations. These stressors contribute to burnout, depression, anxiety, and reduced job satisfaction, all of which may negatively influence patient safety and workforce stability.

Despite the recognized importance of mental health in cardiology, limited data exist from low- and middle-income countries-particularly from Egypt-regarding the concurrent assessment of mental health among both patients and healthcare providers within the same clinical setting.

Therefore, this study aims to estimate the prevalence and correlates of psychiatric symptoms among cardiovascular patients and healthcare providers in a tertiary care center. The results are expected to guide the development of psychosocial support programs and promote mental health awareness in hospital cardiology departments.

Study Design:

Type: Cross-sectional, descriptive, hospital-based study

Setting: Assiut University Heart Hospital

Sample: ~380 cardiovascular patients (systematic random sampling) and all available healthcare providers (census approach)

Tools: Standardized and validated questionnaires including SCL-90R, PSS, PSQI, MBI, and COPE Inventory

Data Analysis: Descriptive and multivariate logistic regression analyses using SPSS v26

ELIGIBILITY:
Inclusion Criteria:

Patients

Age ≥ 18 years. Diagnosed with a cardiovascular disease (e.g., ischemic heart disease, heart failure, valvular disease).

Able to understand and complete self-administered questionnaires or participate in structured interviews.

Provided informed written consent.

Healthcare Providers

Physicians, residents, nurses, or allied staff working in the Department of Cardiovascular Medicine for ≥6 months.

Provided informed written consent.

Exclusion Criteria:

Severe cognitive impairment or communication difficulties that prevent questionnaire completion.

Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with cardiovascular diseases admitted to or attending the outpatient clinics of the Cardiology Department at Assiut University Heart Hospital, and healthcare providers (physicians, residents, nurses, and technicians) currently working in the same department.
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Measuring the prevalence of depressive symptoms among cardiovascular patients assessed by SCL-90R | Within 12 months
  The Symptom Checklist-90-Revised (SCL-90R) will be used to assess depression subscale scores among patients with cardiovascular diseases. A predefined cutoff score indicates the presence of depressive symptoms.
  Unit of measure: Percentage of participants with depressive symptoms (%)
Measuring the prevalence of anxiety symptoms among cardiovascular patients assessed by SCL-90R | Within 12 months
  Anxiety subscale of SCL-90R will be used to quantify anxiety symptoms in patients.
  Unit of measure : Percentage of participants with anxiety symptoms (%)
Prevalence of burnout among healthcare providers assessed by Maslach Burnout Inventory (MBI) | Within 12 months
  The Maslach Burnout Inventory (MBI) will be used to assess emotional exhaustion, depersonalization, and personal accomplishment among cardiology staff.
  Unit of measure : Percentage of participants meeting burnout criteria (%)

SECONDARY OUTCOMES:
Association between sociodemographic and clinical factors and psychiatric symptoms | within 12 months
  Multivariate logistic regression will be used to identify predictors (e.g., age, sex, job type, disease severity) associated with depression, anxiety, and burnout.
  Unit is Odds ratio (95% CI).
Mean Perceived Stress Scale (PSS) score among patients and providers | within 12 months
  Perceived Stress Scale will be used to measure stress levels; higher scores indicate greater perceived stress.
  Unit of measure : Mean PSS score (0-40)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mohammed Tohamy, Ass. Professor, Study Director — Assiut University; Ayman Khairy Hassan, Professor, Study Director — Assiut University; Hossam Loly Abdullah, bachelor's, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Shanafelt TD, Boone S, Tan L, Dyrbye LN, Sotile W, Satele D, West CP, Sloan J, Oreskovich MR. Burnout and satisfaction with work-life balance among US physicians relative to the general US population. Arch Intern Med. 2012 Oct 8;172(18):1377-85. doi: 10.1001/archinternmed.2012.3199. PMID 22911330
- [Result] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Result] Lichtman JH, Froelicher ES, Blumenthal JA, Carney RM, Doering LV, Frasure-Smith N, Freedland KE, Jaffe AS, Leifheit-Limson EC, Sheps DS, Vaccarino V, Wulsin L; American Heart Association Statistics Committee of the Council on Epidemiology and Prevention and the Council on Cardiovascular and Stroke Nursing. Depression as a risk factor for poor prognosis among patients with acute coronary syndrome: systematic review and recommendations: a scientific statement from the American Heart Association. Circulation. 2014 Mar 25;129(12):1350-69. doi: 10.1161/CIR.0000000000000019. Epub 2014 Feb 24. PMID 24566200